CLINICAL TRIAL: NCT03115047
Title: Traitement Des Frissons Lors de la césarienne Sous anesthésie péridurale Durant le Travail - un Essai Clinique randomisé Comparant la dexmédétomidine et la mépéridine
Brief Title: Shivering Treatment After Cesarean Delivery: Meperidine vs. Dexmedetomidine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-7124
Record Dates: First submitted 2017-04-08; First posted 2017-04-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Dexmedetomidine; Meperidine

STUDY DESIGN:
Intervention Model Description: Comparing two groups: experimental (dexmedetomidine) versus control (meperidine)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded randomized study: meperidine and dexmedetomidine will be prepared at the hospital pharmacy in a 10 mL seringue with equivalent dilution in order to gave mL/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine (Experimental): Unique dose of dexmedetomidine injection:
  * intravenous injection
  * 0.35 mcg/kg
  * in two minutes
  * if shivering 5 minutes after delivery
  Interventions: Drug: Dexmedetomidine Injection
- meperidine (Active Comparator): Unique dose of meperidine injection:
  * intravenous injection
  * 0.35 mg/kg
  * in two minutes
  * if shivering 5 minutes after delivery
  Interventions: Drug: Meperidine Injection

INTERVENTIONS:
Drug: Dexmedetomidine Injection — 0.35 mcg/kg intravenous in 2 minutes if shivering 5 minutes after delivery
  Other Names: precedex
  Arms: dexmedetomidine
Drug: Meperidine Injection — 0.35 mg/kg intravenous in 2 minutes if shivering 5 minutes after delivery
  Other Names: demerol
  Arms: meperidine

SUMMARY:
Comparing two treatments for shivering after cesarean delivery for labor dystocia under epidural anesthesia.

DETAILED DESCRIPTION:
It is a double blinded randomized control trial.

Study population: parturients undergoing a cesarean delivery for labor dystocia under epidural anesthesia experiencing shivering grade III or IV on the standardized shivering scale of Crossley and Mahajan

Experimental group: dexmedetomidine 0.35 mcg/kg IV in 2 minutes

Control group: meperidine 0.35 mg/kg IV in 2 minutes

Primary outcome : Time to stop level III and IV shivering on the Crossley and Mahajan standardized shivering scale after the administration of the study drug

Secondary outcome: Response rate, incidence of nausea, vomiting, hypotension, bradycardia, maternal satisfaction and a cost-benefit analysis.

The hypothesis is that dexmedetomidine will act faster, will have a superior response rate with less adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Term > 37 weeks
* American Society of Anesthesiologists Physical Status (ASA PS) I, II
* Weight < 115 kg
* Functional epidural in situ
* In labor requiring cesarean delivery
* Class III or IV shivering on the Crossley and Mahajan standardized shivering scale between five minutes after the baby's birth to the end of the cesarean section

Exclusion Criteria:

* Refusal of the patient and/or the anesthesiologist
* Misunderstanding of the protocol
* Known allergy or contraindication to one of the study drugs
* Emergency cesarean delivery
* American Society of Anesthesiologists Physical Status III, IV, V
* Severe heart, liver or kidney disease,
* Preeclampsia
* Patient taking monoamine oxydase inhibitors
* Sleep apnea
* General anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Parturient, after cesarean delivery
Enrollment: 80 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Stop time | 15 minutes
  Time to stop class III or IV shivering on the Crossley and Mahajan standardized shivering scale after the administration of the study drug (meperidine versus dexmedetomidine)

SECONDARY OUTCOMES:
incidence of adverse effects | 24 hours
  sedation, nausea, vomiting, hypotension and bradycardia
maternal satisfaction | at 24 hours
  satisfaction (yes or no) regarding experience with study drug
response rate | 15 minutes
  percentage of patient responding when the drug is given
cost benefice analysis | 24 hours
  comparing cost of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lavoie, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowley LJ, Buggy DJ. Shivering and neuraxial anesthesia. Reg Anesth Pain Med. 2008 May-Jun;33(3):241-52. doi: 10.1016/j.rapm.2007.11.006. PMID 18433676
- [Background] De Witte J, Sessler DI. Perioperative shivering: physiology and pharmacology. Anesthesiology. 2002 Feb;96(2):467-84. doi: 10.1097/00000542-200202000-00036. No abstract available. PMID 11818783
- [Background] Kranke P, Eberhart LH, Roewer N, Tramer MR. Pharmacological treatment of postoperative shivering: a quantitative systematic review of randomized controlled trials. Anesth Analg. 2002 Feb;94(2):453-60, table of contents. doi: 10.1097/00000539-200202000-00043. PMID 11812718
- [Background] Abdel-Ghaffar HS, Mohamed SA, Fares KM, Osman MA. Safety and Efficacy of Dexmedetomidine in Treating Post Spinal Anesthesia Shivering: A Randomized Clinically Controlled Dose-Finding Trial. Pain Physician. 2016 May;19(4):243-53. PMID 27228512
- [Background] Tsai YC, Chu KS. A comparison of tramadol, amitriptyline, and meperidine for postepidural anesthetic shivering in parturients. Anesth Analg. 2001 Nov;93(5):1288-92. doi: 10.1097/00000539-200111000-00052. PMID 11682416
- [Background] Mittal G, Gupta K, Katyal S, Kaushal S. Randomised double-blind comparative study of dexmedetomidine and tramadol for post-spinal anaesthesia shivering. Indian J Anaesth. 2014 May;58(3):257-62. doi: 10.4103/0019-5049.135031. PMID 25024466
- [Background] Saito T, Sessler DI, Fujita K, Ooi Y, Jeffrey R. Thermoregulatory effects of spinal and epidural anesthesia during cesarean delivery. Reg Anesth Pain Med. 1998 Jul-Aug;23(4):418-23. doi: 10.1016/s1098-7339(98)90017-7. PMID 9690596
- [Background] Crossley AW, Mahajan RP. The intensity of postoperative shivering is unrelated to axillary temperature. Anaesthesia. 1994 Mar;49(3):205-7. doi: 10.1111/j.1365-2044.1994.tb03422.x. PMID 8147511